CLINICAL TRIAL: NCT05853146
Title: Fetal Heart Rate Characterization Using Innovative Advanced Non-invasive Technology
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oxitone Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 0262-22
Record Dates: First submitted 2023-04-23; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Fetus Pulse Monitoring
Keywords: fetus; pulse; monitoring; pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- pregnant women: Healthy women in their third trimester of pregnancy with one fetus
  Interventions: Device: Oxitone 1000M

INTERVENTIONS:
Device: Oxitone 1000M — World's First FDA-cleared Wrist-Sensor Pulse Oximetry Monitor

SUMMARY:
The purpose of the study is to examine the effectiveness and reliability of fetal heart rate monitoring by the Oxitone device.

Today, fetal monitoring is carried out with an external approach using a Doppler transducer placed on the mother's abdomen or with an internal approach only after water breaks and during active labor by connecting an electrode to the head of the fetus.

Oxyton's technology collects various physiological indicators and calculates an estimation of the fetal pulse. This monitoring method has a wide potential for use as part of pregnancy monitoring and perhaps even during childbirth.

Fetal heart rate will be measured in pregnant women in the third trimester of pregnancy with one fetus. The patients will wear the Oxitone device at the same time as Doppler monitoring in the hospital. An analysis of the data will be performed in comparison to the current accepted fetal monitor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the age of 18-50

Exclusion Criteria:

* Clotting disorders, diabetes, currently taking psychotropic medications

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women in the third trimester of pregnancy with one fetus.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
fetus pulse | through study completion, an average of 1 year
  fetus pulse calculated by a new algorithm